CLINICAL TRIAL: NCT01638351
Title: Effects of Resistance Training on Muscle Dysfunction in Elderly Patients With Type 2 Diabetes Mellitus
Brief Title: Resistance Training in Diabetic Elder Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201110029RC
Record Dates: First submitted 2012-07-08; First posted 2012-07-11 (Estimated); Last update posted 2012-11-16 (Estimated); Status verified 2012-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes mellitus; Resistance exercise; Elderly; Skeletal muscle dysfunction; Metabolomics
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (Active Comparator): Participants in this arm will receive a brochure specific for type 2 diabetes mellitus about the general principles of exercise, nutrition, and diet. They are asked to maintain their activity level.
  Interventions: Behavioral: Usual care
- Resistance exercise (Experimental): Progressive resistance training, 3 times a week for 12 weeks
  Interventions: Behavioral: Resistance exercise

INTERVENTIONS:
Behavioral: Resistance exercise — Progressive resistance exercise training, 3 times a week for 12 weeks.
  Arms: Resistance exercise
Behavioral: Usual care — Participants in this arm will receive a brochure specific for type 2 diabetes mellitus about the general principles of exercise, nutrition, and diet. They are asked to maintain their activity level.
  Arms: Usual care

SUMMARY:
The purpose of this study is to investigate the effect of a 12-week progressive resistance training program on the skeletal muscle function, glycemic control, functional capacity, and quality of life in the elderly with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* 65 years old or older
* no clinical diagnosis of cardiovascular disease
* patients with or without type 2 diabetes mellitus

Exclusion Criteria:

* glycated hemoglobin > 10%
* pulmonary disease
* cancer
* cognitive dysfunction
* any neurological or musculoskeletal disease that will affect exercise performance

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 49 (Actual)
Dates: Start 2011-12; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Maximal muscle strength | Twelve weeks
  This outcome measure includes upper and lower body maximal muscle strength.

SECONDARY OUTCOMES:
Physical body function | Twelve weeks
  This outcome will be assessed by one minute sit-to-stand test and timed "Up and Go" test.
Quality of life | Twelve weeks
  This outcome measure will be assessed by the diabetes-specific questionnaire.
Waist circumference | Twelve weeks
Body mass index | Twelve weeks
  This outcome measure includes the measurements of body height and body weight.
Functional capacity | Twelve weeks
  Peak oxygen consumption will be determined by graded exercise test to assess functional capacity.
Blood biochemical parameters | Twevle weeks
  This outcome measure includes the analysis of fasting glucose, glycated hemoglobin, lipid profile, C-reactive protein, and related metabolites.
Muscle oxygenation | Twelve weeks
  Muscle oxygenation will be assessed during exercise

CONTACTS AND LOCATIONS:
Overall Officials: Ying-Tai Wu, Ph.D., Study Chair — School and Graduate Institute of Physical Therapy, College of Medicine, National Taiwan University (R.O.C.)
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Castaneda C, Layne JE, Munoz-Orians L, Gordon PL, Walsmith J, Foldvari M, Roubenoff R, Tucker KL, Nelson ME. A randomized controlled trial of resistance exercise training to improve glycemic control in older adults with type 2 diabetes. Diabetes Care. 2002 Dec;25(12):2335-41. doi: 10.2337/diacare.25.12.2335. PMID 12453982
- [Background] Dunstan DW, Daly RM, Owen N, Jolley D, De Courten M, Shaw J, Zimmet P. High-intensity resistance training improves glycemic control in older patients with type 2 diabetes. Diabetes Care. 2002 Oct;25(10):1729-36. doi: 10.2337/diacare.25.10.1729. PMID 12351469
- [Background] Brandon LJ, Gaasch DA, Boyette LW, Lloyd AM. Effects of long-term resistive training on mobility and strength in older adults with diabetes. J Gerontol A Biol Sci Med Sci. 2003 Aug;58(8):740-5. doi: 10.1093/gerona/58.8.m740. PMID 12902533
- [Background] Cheung NW, Cinnadaio N, Russo M, Marek S. A pilot randomised controlled trial of resistance exercise bands in the management of sedentary subjects with type 2 diabetes. Diabetes Res Clin Pract. 2009 Mar;83(3):e68-71. doi: 10.1016/j.diabres.2008.12.009. Epub 2009 Jan 20. PMID 19157617